CLINICAL TRIAL: NCT00662870
Title: Safety, Immunogenicity and Lot Comparability of DAPTACEL™ (Aventis Pasteur Classic Five-component Pertussis Vaccine in Combination With Tetanus and Diphtheria Toxoids Adsorbed) When Administered With Other Recommended Vaccines at 2, 4, 6, and 15 to 16 Months of Age.
Brief Title: Study of the Safety, Immunogenicity and Lot Comparability of DAPTACEL When Administered With Other Recommended Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P3T06
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Diphtheria; Tetanus; Whooping Cough; Polio; Haemophilus Influenzae Type b
Keywords: DAPTACEL; Diphtheria; Tetanus; Whooping Cough; Polio; Haemophilus influenzae type b; Pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Haemophilus Infections | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Tetanus Toxoid; pentacel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- DAPTACEL Lot 1 (Experimental): Participants receiving Diphtheria and Tetanus Toxoids and Acellular Pertussis vaccine (DAPTACEL) Lot 1
  Interventions: Biological: DAPTACEL® (Diphtheria and Tetanus Toxoids and Acellular Pertussis vaccine)
- DAPTACEL Lot 2 (Experimental): Participants receiving Diphtheria and Tetanus Toxoids and Acellular Pertussis vaccine (DAPTACEL) Lot 2
  Interventions: Biological: DAPTACEL® (Diphtheria and Tetanus Toxoids and Acellular Pertussis vaccine)
- DAPTACEL Lot 3 (Experimental): Participants receiving Diphtheria and Tetanus Toxoids and Acellular Pertussis vaccine (DAPTACEL) Lot 3
  Interventions: Biological: DAPTACEL® (Diphtheria and Tetanus Toxoids and Acellular Pertussis vaccine)
- Pentacel (Active Comparator): Participants receiving Pentacel vaccine
  Interventions: Biological: Pentacel: DTaP-IPV/Hib

INTERVENTIONS:
Biological: DAPTACEL® (Diphtheria and Tetanus Toxoids and Acellular Pertussis vaccine) — 0.5 mL, Intramuscular
  Other Names: DAPTACEL®
  Arms: DAPTACEL Lot 1; DAPTACEL Lot 2; DAPTACEL Lot 3
Biological: Pentacel: DTaP-IPV/Hib — 0.5 mL, Intramuscular
  Other Names: Pentacel
  Arms: Pentacel

SUMMARY:
This study was designed to assess the lot comparability of DAPTACEL, as well as the safety and immunogenicity of DAPTACEL when co-administered with other recommended infant vaccines.

Stage I Primary Objectives:

1. To assess the lot-comparability of immunogenicity of DAPTACEL by when co-administered with other recommended vaccines.
2. To compare the immune response to DTaP-IPV/Hib (Pentacel) with those of three lots of DAPTACEL when co-administered with other recommended vaccines.
3. To compare the immune response of PRP-T antigen in Pentacel with that of ActHIB concurrently administered in a different injection site with DAPTACEL when these vaccines are co-administered with other recommended vaccines.

Stage II Primary Objectives:

1. To compare the immune response of DAPTACEL when the 4th dose is co-administered with Hib or other infant vaccines.
2. To compare the the immune response of Pentacel with those elicited by DAPTACEL when co-administered with ActHIB in toddlers.

DETAILED DESCRIPTION:
This is a two-stage, randomized, multi-center study to assess the safety, immunogenicity and lot comparability of DAPTACEL

ELIGIBILITY:
Inclusion Criteria :

* Healthy infants 2 months of age.
* Infants with at least 37 weeks of gestation at delivery.
* Signed informed consent from parent or guardian.
* Able to attend the scheduled visits and to comply with the study procedure.
* Subjects must have received the first dose of hepatitis B vaccine from birth to 28 days prior to the first dose of DAPTACEL or Pentacel.

Exclusion Criteria :

* Clinically significant findings on review of systems or physical examination (determined by investigator or sub-investigator to be sufficient for exclusion).
* Known or suspected hypersensitivity to any component of the study vaccine to be administered.
* Known or suspected impairment of immunologic function or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Known HIV-positive mother.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay or neurologic disorders.
* Chronic medical, congenital, developmental or surgical disease.
* Participation in any other experimental vaccine trial.
* Any condition which, in the opinion of the investigator or sub-investigator, would interfere with the evaluation of the vaccine or pose a health risk to the subject.
* Prior history of having received more than one dose of hepatitis B vaccine, any diphtheria, tetanus and acellular pertussis combination vaccine (DTaP), diphtheria, tetanus and whole-cell pertussis combination vaccine (DTwP), Haemophilus influenzae type b (Hib)-conjugate vaccine, poliovirus vaccine or pneumococcal conjugate vaccine

Ages: 42 Days to 84 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1941 (Actual)
Dates: Start 2001-05; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immune response of DAPTACEL after vaccination. | 30 days post-vaccination 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur, Inc.
Locations (26):
- United States (26):
  - Fayetteville, AR 72703, Arkansas
  - Jonesboro, AR 72401, Arkansas
  - Little Rock, AR 72211, Arkansas
  - Fountain Valley, CA 92708, California
  - Englewood, CO 80112, Colorado
  - Norwich, CT 06360, Connecticut
  - Orlando, FL 32856, Florida
  - Marietta, GA 30062, Georgia
  - Chicago, IL 60614, Illinois
  - Bardstown, KY 40004, Kentucky
  - Bossier City, LA 71111, Louisiana
  - Bridgeton, MO 63044, Missouri
  - Rochester, NY 14620, New York
  - Chapel Hill, NC 27514, North Carolina
  - Portland, OR 97201, Oregon
  - Norristown, PA 19401, Pennsylvania
  - Pittsburgh, PA 15213, Pennsylvania
  - Pittsburgh, PA 15241, Pennsylvania
  - Kingsport, TN 37664, Tennessee
  - Austin, TX 78758, Texas
  - Fort Worth, TX 76107, Texas
  - San Antonio, TX 78205, Texas
  - Provo, UT 84604, Utah
  - Spokane, WA 99220, Washington
  - LaCrosse, WI 54601, Wisconsin
  - Marshfield, WI 54449, Wisconsin

REFERENCES:
- [Result] Guerra FA, Blatter MM, Greenberg DP, Pichichero M, Noriega FR; Pentacel Study Group. Safety and immunogenicity of a pentavalent vaccine compared with separate administration of licensed equivalent vaccines in US infants and toddlers and persistence of antibodies before a preschool booster dose: a randomized, clinical trial. Pediatrics. 2009 Jan;123(1):301-12. doi: 10.1542/peds.2007-3317. PMID 19117896
- See also: Related Info — http://www.sanofipasteur.com